CLINICAL TRIAL: NCT00701259
Title: A Phase III, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Trial of Fourteen Day Treatment With Lansoprazole 15 mg or 30 mg Once a Day in Frequent Nighttime Heartburn
Brief Title: Efficacy/Safety of Lansoprazole in Patients With Frequent Nighttime Heartburn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Regulatory Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRSW-GN-305
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Frequent Heartburn
Keywords: Frequent heartburn, proton pump inhibitor, lansoprazole; Treatment of; over 14 days
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 15 mg lansoprazole
  Interventions: Drug: Lansoprazole
- 2 (Experimental): 30 mg lansoprazole
  Interventions: Drug: Lansoprazole
- 3 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole 15 mg once per day for 14 days
  Other Names: Prevacid - United States
  Arms: 1
Drug: Lansoprazole — Lansoprazole 30 mg once per day for 14 days
  Arms: 2
Drug: placebo
  Arms: 3

SUMMARY:
Heartburn, a burning sensation in the chest or throat, occurs in many individuals when acidic stomach contents move upward into the esophagus from the stomach. This study will investigate the safety and efficacy of lansoprazole 15 mg or 30 mg administered once a day in preventing frequent nighttime heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing heartburn at least 2 days per week during the nighttime period over the past month.
* Having heartburn that responds to heartburn medication.
* Be willing to discontinue the use of heartburn treatment for 7 days prior to inclusion in the study.

Exclusion Criteria:

* Having history of erosive esophagitis or gastroesophageal reflux disease diagnosed by a physician and confirmed by testing (endoscopy).
* Be unwilling to take only the study medication, and antacid provided as a rescue medication for relief of acute heartburn during the study.

"Other protocol-defined inclusion/exclusion criteria may apply"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Actual)
Dates: Start 2007-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Percentage of nighttimes with no heartburn during 14 days of double-blind treatment in subjects with frequent heartburn. | 14 days

SECONDARY OUTCOMES:
Proportion of 24 hour days with no heartburn during 14 days of treatment. Proportion of subjects with no heartburn during day 1 (the 24 hours following the first dose. The evaluation of lansoprazole safety. | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Not applicable - enrollment complete, Parsippany, New Jersey, United States